CLINICAL TRIAL: NCT01764763
Title: Intraoperative Epiaortic Scanning for Preventing Early Stroke After Off-pump Coronary Artery Bypass
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2010-0868
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non epiaortic group: non epiaortic group ( n=1019)
- epiaortic group: epiaortic group ( n=1273)

SUMMARY:
Recently epiaortic ultrasound scanning (EAS) has been recommended as an intraoperative tool to accurately assess ascending aorta disease. To date, several studies have reported that EAS is superior to TEE and surgical palpation

ELIGIBILITY:
Inclusion Criteria:

patients underwent who isolated off-pump coronary artery bypass

Exclusion Criteria:

1. combined carotid procedures
2. preoperative cerebral haemorrhage
3. nonoperative unstable vital signs such as ventricular fibrillation or cardiac arrest

Ages: 31 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2001 to December 2011, 2292 patients who underwent isolated off-pump coronary artery bypass at Yonsei Cardiovascular Hospital in Seoul
Sampling Method: Non-Probability Sample
Enrollment: 2292 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Early Stroke After Off-pump Coronary Artery Bypass | number of incidence of early strok from surgery to discharge, an expected average of 5 weeks